

Study protocol December 1, 2017

UIC PAF #: 2014-01275

UIC IRB protocol #: 2014-1214

Clinicaltrials.gov registration #: NCT02319967

Patient-Centered Outcomes Research Institute, contract # AS 1307-05420

Project period: March 1, 2014 – May 31, 2017

### TABLE OF CONTENTS

| | | Page |
|---|---|---|
| I. | Executive summary | 3 |
| II. | Overview of pragmatic trial | 4 |
| III. | Primary and secondary aims | 4 |
| IV. | Study population | 4<br>5 |
| V. | Interventions and comparators | 7 |
| VI. | Randomization | 9 |
| VII. | Data collection | 9 |
| | A. Screening and enrollment (registration) into the study (in person) | |
| | B. 1-month follow-up visit after ED discharge (telephone) | |
| | C. 3-month follow-up visit after ED discharge (telephone) | |
| | D. 6-month follow-up visit after ED discharge (in person) | |
| | E. 12-month follow-up visit after ED discharge (telephone) | |
| VIII. | Outcomes | 10 |
| | A. Primary outcomes | |
| | B. Secondary outcomes | |
| IX. | Analysis plan | 11 |
| X. | Barriers and facilitators of successfully implementing the intervention | 13 |
| | (secondary aim) | |
| XI. | Timeline / milestones | 14 |
| XII. | Protection of human subjects | 15 |
| | A. Risks to human subjects | |
| | B. Source of materials | |
| | C. Potential risks | |
| | D. Adequacy of protection against risks | |
| | E. Potential benefits of the proposed research to the subjects and others | |
| | F. Importance of the knowledge to be gained | |
| | G. Data safety monitoring plan | |
| | H. Clinicaltrials.gov requirements | |
| | I. Inclusion of women and minorities | |
| XIII. | References | 19 |
| XIV. | Appendices | 24 |
| | A. CAPE tool | |
| | B. Outline of home visit procedures | |

#### I. Executive summary

1 2

Chicago is an epicenter for asthma health disparities in the United States, with African American 3 4 children 5-11 years old bearing a disproportionate share of the burden. Gaps in implementation at provider and patient levels contribute to these asthma disparities, with studies suggesting that 5 minority children are less likely than white children to be prescribed and use guideline-6 7 recommended asthma care, respectively. Effective strategies to implement national asthma 8 guideline recommendations in this population are needed. As part of a Patient-Centered Outcomes Research Institute contract (AS 1307-05420; Coordinated Healthcare Interventions for Childhood 9 Asthma Gaps in Outcomes [CHICAGO] Plan), we used methods in user-centered design to inform 10 the development of interventions to implement asthma guidelines in the ED and at home. We then 11 conducted a pragmatic trial to evaluate the effectiveness of ED and home-based interventions on 12 patient- and caregiver-centered endpoints. 13

#### II. Overview of the pragmatic trial

15 16

- The CHICAGO Plan was a randomized 3-arm parallel group, multi-center pragmatic trial in six 17
- 18 Emergency Departments (EDs) affiliated with public or private hospitals who served a high
- proportion of black or Latino children in Chicago to compare: 1) an ED-only intervention 2) an 19
- ED-plus-home intervention; and 3) Enhanced usual care. Eligibility criteria were intended to be 20
- clinically applicable and recruitment took place in multiple EDs serving underserved communities 21
- in Chicago (six Clinical Centers serving different populations of children 5-11 years presenting 22
- with asthma). Data collection employed validated approaches, but were also intended to minimize 23 24

participant burden

25 26

#### III. Primary and secondary aims

27

- 28 Primary aim
- Conduct a 3-arm multi-center pragmatic trial comparing the effectiveness of the ED-only, ED-29 plus-home, and usual care strategies. 30

31 32

33

34

- Secondary aims
  - Examine the potential for heterogeneity of treatment effects.
  - Identify barriers and facilitators of successfully implementing the interventions to inform subsequent research to accelerate the uptake of study findings.

#### **Outcomes assessments**



#### Intervention



<u>Figure 1</u>: Children ages 5 to 11 years who presented with uncontrolled asthma to the emergency department (ED) were randomly allocated to one of three groups: Enhanced usual care vs. ED-based intervention using the CHICAGO Action Plan after Emergency department discharge (CAPE) decision support and communication tool for children and caregivers (ED-only), vs. the same ED-only intervention plus community health worker-led home visits at 2-3 days, 2 weeks, 1 month, 3 months, and 6 months after ED discharge to help implement the CAPE and reduce environmental triggers (ED-plus-home). Outcomes were assessed at baseline (in-person prior to ED discharge), 1 month (via phone), 3 months (via phone), and 6 months (in-home or via phone; time point for the primary outcome) after ED discharge.

#### IV. Study population

Eligibility criteria were designed to be clinically relevant and feasible to implement in an ED setting. Due to lower than expected randomizations during the first half of the recruitment period, we modified the study eligibility criteria after review by an independent Data and Safety and Monitoring Board, institutional IRBs (Site-specific IRB approval dates: Lurie – 9/14/2015; Rush – 9/8/2015; Sinai – 9/10/2015; Stroger – 8/18/2015; UC – 9/1/2015; UIC – 7/28/2015), and discussions with the program officer from the Patient-Centered Outcomes Research Institute. Original and revised eligibility criteria are below; to be eligible, patients needed to meet all inclusion criteria and none of the exclusion criteria below.

#### **ORIGINAL ELIGIBILITY CRITERIA:**

Original eligibility criteria approved by prime site IRB (UIC #2014-1214) on 12/19/2014.

#### **Inclusion criteria (all of the following):**

- 1. Child is 5-11 years of age (a population in whom a diagnosis of asthma is generally reliable, and in whom exacerbations are common);
  - 2. Child is presenting to the ED, urgent care center, or observation unit at a participating clinical center (Anne and Robert H. Lurie Children's Hospital of Chicago, Sinai Health System's Mount Sinai Hospital, John H. Stroger Jr. Hospital of Cook County Health & Hospitals System, Rush University Medical Center, University of Chicago Medicine Comer Children's Hospital, and the University of Illinois Hospital & Health Sciences System);
- 70 3. Child is treated with at least 1 dose of an inhaled or nebulized short-acting bronchodilator (quick-relief medication);
  - 4. Child received systemic corticosteroids in the ED;
- Child and caregiver approached at least 1 hour after receipt of the first dose of quick-relief
   medication or systemic corticosteroids, whichever occurred last;
  - 6. Diagnosis of asthma exacerbation by treating clinician;
  - 7. Treating ED clinician indicates the child is likely to be discharged to home;
  - 8. Caregiver reports that English or Spanish is the preferred language at home.

#### **Exclusion criteria (none of the following):**

- 1. Caregiver declines to provide informed consent, or the child declines to provide assent;
- 2. Child is discharged to a location other than home (e.g., hospital or another healthcare facility);
- 3. Child or another member of the child's primary household is a current or previous participant in the CHICAGO Plan;
- 4. Child is enrolled in another study involving a health-related intervention;
- 5. A CHW is already visiting the home as part of another program;
- 86 6. Child is expected to move out of Chicago within the next 6 months.

87 88

89

90

62

65

66

67

68

69

72

75

76

77 78 79

80

#### **REVISED ELIGIBILITY CRITERIA:**

Revised eligibility criteria approved by prime site IRB (UIC #2014-1214) on 7/28/2015. Revisions occurred over a period of a few months across all of the other clinical centers (after local institutional review).

91 92 93

94 95

96

97

98

99

100

#### **Inclusion criteria (all of the following):**

- 1. Child is 5-11 years of age (a population in whom a diagnosis of asthma is generally reliable, and in whom exacerbations are common);
- 2. Child is presenting to the ED, urgent care center, or observation unit at a participating clinical center (Anne and Robert H. Lurie Children's Hospital of Chicago, Sinai Health System's Mount Sinai Hospital, John H. Stroger Jr. Hospital of Cook County Health & Hospitals System, Rush University Medical Center, University of Chicago Medicine Comer Children's Hospital, and the University of Illinois Hospital & Health Sciences System);
- 101 3. Child is treated with at least 1 dose of an inhaled or nebulized short-acting bronchodilator (quick-relief medication);
- 4. Child received systemic corticosteroids in the ED OR the caregiver reported at least 1
   additional acute care visit for asthma in the previous 6 months (defined as an asthma-related
   ED visit or urgent care visit, or course of systemic corticosteroids);
- 5. Child and caregiver approached at least 1 hour after receipt of the first dose of quick-relief medication or systemic corticosteroids, whichever occurred first;

- 108 6. Diagnosis of asthma exacerbation by treating clinician;
- 7. Treating ED clinician indicates the child is likely to be discharged to home;
- 8. Caregiver reports that English or Spanish is the preferred language at home.

#### 

#### **Exclusion criteria (none of the following):**

- 1. Caregiver declines to provide informed consent, or the child declines to provide assent;
- 2. Child is admitted to an intensive care unit or transferred to another healthcare facility;
- 3. Child or another member of the child's primary household is a current or previous participant in the CHICAGO Plan;
- 4. Child is enrolled in another study involving a health-related intervention;
- 5. A Community Health Worker (CHW) is already visiting the home as part of another program;
- 119 6. Child does not reside in Chicago.

#### V. Interventions and comparators

All children who participated in the CHICAGO Plan received asthma care per their ED clinicians. In addition, the CHICAGO Plan's ED Coordinator provided all participants two metered dose inhaler (MDI) spacers free-of-charge and used teach-to-goal methodology (repeated rounds of education and evaluation until the child achieves mastery) to educate the child and the caregiver about appropriate MDI inhaler technique. Patient education regarding the MDI device was selected because it is commonly used for quick-relief medications and is also the device for many inhaled controller medications. Children were then randomly assigned to either of two active comparators or enhanced usual care.

1. ED-only. Based on feedback from our stakeholders, we developed the CHICAGO Action Plan after Emergency department discharge tool (CAPE; APPENDIX A1); a culturally tailored and literacy-appropriate communication tool for use on ED discharge. Based on the ED treating clinician's discharge instructions, a CHICAGO Plan ED Coordinator utilized the CAPE to support guideline recommended asthma care on ED discharge (a course of systemic corticosteroids; daily inhaled corticosteroids or other controller; as needed quick-relief inhaled medication; education about the medications and appropriate inhaler technique; education about asthma trigger avoidance; and a post-discharge follow-up appointment) and to support appropriate asthma self-management in the home. The CAPE tool uses simplified language, visual learning, and options for individualization to facilitate communication about discharge instructions between clinicians and the child and caregiver.

2. ED-plus-home. Participants randomly allocated to the ED-plus-home intervention received the same ED-only intervention described above but were also offered up to five home visits over 6 months conducted by a CHW visits to: 1) assist in the implementation of the ED discharge instructions, 2) update the asthma treatment plan with input from the patient's ambulatory clinician utilizing the CAPE tool called the Asthma Home Plan (APPENDIX A2), 3) develop a plan to manage asthma during school hours (e.g., access to quick-relief medications, action plan in case of respiratory difficulty), and 4) develop a specific and feasible plan to reduce environmental triggers at home (e.g., environmental tobacco smoke, roach, mice). Home visits were scheduled for 60 to 90 minutes, and occurred

- approximately at 2-3 days, 2 weeks (14 days), 1 month (30 days), 3 month (90 days), and 6 months (180 days) after ED discharge.
- 3. Enhanced usual care. Based on stakeholder feedback, we modified usual care so that 157 children in the "usual care" group also received teaching about appropriate MDI technique 158 using teach-to-goal methodology and two MDI spacers free-of-charge, as well as doorknob 159 hangers depicting facts about asthma unrelated to the study interventions. We therefore 160 refer to this group as "Enhanced usual care." To describe usual care at each site, the site 161 project manager conducted chart abstractions (masked to treatment assignment). Site 162 project managers were to complete chart abstractions within 3 business days of enrolling 163 the participant in the study. 164

154

155156

#### VI. Randomization

Randomization occurred at the patient level, with permuted block sizes stratified by site and race (black vs. non-black). Based on data from the Clinical Centers, we expected about 70% of enrolled participants to be black, 23% to be white, and that the remainder would be mostly Asian. Of the planned enrollment of 640 children, we expected 15% to be Hispanic/Latino. Stratification by race for the purposes of randomization was "Black" (those who selected Black or African American, includes multi-race if at least one race was Black or African American) vs. "non-Black" (American Indian/Alaskan Native, Asian, Native Hawaiian or other Pacific Islander, white, and multi-race if none are Black or African American).

The CHICAGO Plan Research Electronic Data Capture (REDCap) system for study personnel (available 24 hours x7 days/week) provided the random treatment assignment: ED-only, ED-plushome, or Enhanced usual care.

#### VII. Data collection

A. Screening and enrollment (registration) into the study (in person; ~40 minutes). The ED coordinator, a member of the research team, at each Clinical Center screened patients in the ED, Urgent Care, or Observation Unit after treatment initiation for asthma exacerbation and before discharge. The ED coordinator obtained verbal assent from the ED clinician prior to approaching the child/caregiver for informed consent. Following informed consent, the ED coordinator obtained Baseline data, registered the patient in a customized, secure, on-line CHICAGO Plan REDCap portal developed by the DCC, then obtained the treatment assignment (ED-only, ED-plus-home, or Enhanced usual care). The ED Coordinator offered to arrange the date/time of the 1-month follow-up visit (see below).

B. 1-month follow-up contact after discharge (telephone; ~15 minutes). Post-baseline data collection was performed by the DCC Research Assistant, who was masked to treatment assignment. The Research Assistant conducted a telephone interview to assess outcomes approximately 1 month after discharge. The interview was also designed to collect / update contact information and to promote retention in the CHICAGO Plan. The DCC Research Assistant arranged date/time of the 3-month follow-up visit (see below), or inquired about the best time to call again.

C. 3-month follow-up contact after ED discharge (telephone; ~15 minutes). The DCC Research Assistant, masked to treatment assignment, conducted a telephone interview to assess outcomes approximately 3 months after ED discharge. The interview was also designed to collect / update contact information and to promote retention in the CHICAGO Plan. The DCC Research Assistant arranged date/time of the 6-month follow-up visit (see below), or inquired about the best time to call again.

D. 6-month follow-up contact after discharge (in person or by telephone; ~40 minutes). The DCC Research Assistant, masked to treatment assignment, conducted a study visit in person or via telephone (per participant preference) to assess outcomes approximately 6 months after discharge. The in-person visit afforded the ability to conduct an assessment of home trigger avoidance;

review inhaler technique; and assess cACT (child) and PACQLQ, which are more easily collected 212 during in-person visits. 213

214 215

216

217

218

E. 12-month follow-up contact after discharge (in person or by telephone; ~40 minutes). We proposed re-assessing outcomes at 12 months to examine the durability of effects observed at 6 months. Despite significant efforts, retention in the study also proved to be challenging, and therefore the 12-month follow-up visit was discontinued at the request of PCORI in September 2016.

219 220 221

#### **VIII. Outcomes**

222 223

224

225

226

227

228

229

230 231 The selection of primary outcomes was based on several criteria: 1) patient-centeredness, defined as domains identified as important by children and their caregivers; as described in our previous publications; 2) availability of validated measures in English and in Spanish that could be administered in person and by phone; 3) plausibility that such measures could be responsive to an effective intervention in the target population; and 4) limited burden (e.g., time) for study participants. On this basis, we selected two NIH Patient-Reported Outcomes Measurement Information System (PROMIS) measures as primary outcomes (1 for the child and 1 for the caregiver). Several measures were selected for secondary outcomes to address recommendations of national asthma guidelines, expressed preferences of caregivers and other stakeholders, and to compare results of the CHICAGO Plan with previous studies.

232 233 234

235

236

237

238

#### A. Primary outcomes

1. The change in asthma impact at 6 months compared to the baseline assessed in the ED served as the primary outcome in children. In children 5 to 7 years, we assessed asthma impact using the PROMIS Parent Proxy Short Form v1.0 – Asthma Impact 8a. In children 8 to 11 years, we used the PROMIS Pediatric Short Form v1.0 – Asthma Impact 8a.

239 240

2. The change in Satisfaction with Participation in Social Roles at 6 months compared to the baseline assessed in the ED served as the primary outcome in the caregiver. We used the PROMIS Short Form v1.0 – Satisfaction with Participation in Social Roles 4a.

242 243 244

246

247

248

241

#### B. Secondary outcomes

For children: 245

- 1) The Childhood Asthma Control Test (cACT) at 6 months compared to the baseline assessed in the ED
- 2) Acute care visits at 6 months (number of all-cause urgent care visits, ED visits, hospitalizations, using electronic health records)

compared to the baseline assessed in the ED

249 250 251

#### For caregivers:

252 253 254

1) Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) at 6 months compared to the baseline assessed in the ED 2) NIH PROMIS measures for anxiety, depression, fatigue, sleep disturbance at 6 months

255

256

- 258 Indicators of guideline-consistent asthma care provided on ED discharge:
- 1) Systemic corticosteroids prescribed for use at home (yes/no)
- 260 2) Inhaled corticosteroids or another controller medication prescribed for use at home (yes/no)
  - 3) Quick-relief medications prescribed for use at home (yes/no)
    - 4) Follow-up appointment scheduled (yes/no)
  - Child's/caregiver's self-management practices after ED discharge:
    - 1) Filled prescriptions for systemic corticosteroids within 7 days of ED discharge (yes/no)
    - 2) Filled prescription for inhaled corticosteroids or other asthma controller within 7 days of ED discharge (yes/no)
    - 3) Attendance at outpatient appointment with patient-identified asthma provider within 4 weeks of ED discharge (yes/no)

#### IX. Analysis plan

All randomized subjects were included in the primary analysis, unless subjects were terminated due to ineligibility. Baseline sociodemographic and clinical characteristics in the intervention and control groups were compared using the frequency and percentages for categorical variables and median with inter-quartile or mean with standard error for continuous variables. For bivariate analyses, the pairwise comparisons between three intervention arms for the change in primary and some secondary outcomes from baseline to 3 or 6 months were tested by Wilcoxon rank sum test. The W statistic, p-value and mean rank were reported together with horizontal mirror bar plots. For primary outcomes, a statistical significance occurred when p-value was less than 0.0167 after Bonferroni correction for three pairwise comparisons (0.05/3). In addition, chi-square tests were also conducted for other secondary outcomes.

To address missing data in the analyses, we checked the missing completely at random (MCAR) assumption and then employed a multiple imputation strategy. Using a logistic regression method described in Hedeker & Gibbons (2006), we found that the current outcome missingness was not statistically associated with previous observed outcomes across time. Additional characteristics comparisons between participants with and without missing primary outcomes across time was also done using Chi-square tests for categorical variables and Mann-Whitney U test for continuous variables. No statistical difference was observed between the two groups (i.e. with and without missing primary outcomes). We therefore used a fully conditional specification (FCS) approach to impute the missing values with variables of interest in the primary analysis models for 30 imputations. The raw and imputed data had similar distributions (mean, standard deviation, minimum and maximum values).

Since the two primary outcomes were not normally distributed and our data satisfied the MCAR assumption, we used generalized estimating equations (GEE) to examine the effect of intervention group on outcomes at 3 and at 6 months compared to that of the enhanced usual care group using ordinal logistic regression models; the continuous dependent variables were categorized into quartiles. The main predictors of the unadjusted GEE models were time (0, 1, 3, and 6 months), intervention group, and their interactions. In an adjusted model, we added pre-specified covariates including, race (Black vs. non-Black), ethnicity (Latino vs. non-Latino), gender (boy vs. girl),

health insurance (Public aid vs. Other), site enrolled (sites 1 to 6), number of all-cause acute care use in the 12 months prior to enrollment (at least one vs. none). To access the intervention effect between groups across time, we reported our results as odds ratios (ORs for higher quartiles) of interactions between study group and time and their 98% confident intervals [CIs; corresponding to a 2-sided alpha=0.0167) to account for Bonferroni adjustments for the three pairwise comparisons.

308 309 310

311

312

313

303 304

305 306

307

In secondary analyses, we explored heterogeneity of treatment effects by adding a three-way interaction between intervention, time, and a subgroup factor in the model described previously. Pre-specified subgroup factors included race (Black vs. non-black), ethnicity (Latino vs. non-Latino), gender (boy vs. girl), and number of all-cause acute care use in the 12 months prior to enrollment (at least one vs. none).

314 315 316

317

318

319

320

321

322

323

324

325

326

327

328

329

330

331

332

333

334

335

<u>Power / sample size calculation.</u> The power analyses did not incorporate adjustment for the presence of two primary outcomes. Such an adjustment is not commonly made in biomedical trials, as multivariate (viz. MANOVA) analyses are not commonly conducted. The power analysis for single outcomes employed the Rochon (1991) method based on Hotelling's T-squared, which was adapted to a 3-group comparison by adjusting the alpha level using a Bonferroni-style technique. This approach tends toward a conservative (larger) sample size. We proposed to enroll and randomize 640 participants over 18 months (~200-215 for each of the 3 treatment groups). Assuming evaluable data in 80% of enrolled participants (n=512) at 6 months (the timepoint for the analyses of the primary outcomes), sample size calculations suggest ample power. Our approach was based on the methods of Rochon, with a Bonferroni adjustment for 3 pair-wise comparisons (2-sided  $\alpha = 0.05/3 = 0.0167$ ; enhanced usual care and two active intervention groups), power 80%, 4 measurements per individual (0, 1, 3, and 6 months), within individual correlation 0.80, correction for within ED clustering (design effect of 2), and a coefficient of determination (R2) for control of individual-level demographics = 0.15. Based on these considerations, a sample size of 426 (well within the expected sample size of 512) was estimated to be sufficient for a minimum detectable difference of 0.35 standard deviations (SDs) (midway between Cohen's "small" (0.2 SDs) and "medium" (0.5 SDs) effect sizes) for each of the two primary continuous outcomes compared pairwise across the three treatment groups. The minimum detectable difference of 0.35 SDs corresponds to sufficient power to detect a T-score difference of 3.5, which is approximately mid-way between estimates of the minimum important difference (MID) for PROMIS T-scores (2 to 5).

#### X. Barriers and facilitators of successfully implementing the intervention (Secondary aim)

Health system interventions are often multi-component, and when they successfully improve care or outcomes, it is helpful to know whether all components of the intervention were necessary for success. Also, when care outcomes are not improved, it is unclear if barriers to implementation (fidelity) or lack of efficacy contributed to a lack of effect. We therefore a mixed -methods approach to 1) assess the fidelity of implementing the ED-only and ED-plus-home interventions; and 2) conduct interviews to debrief with study staff and a convenience sample of caregivers.

- (1) Intervention fidelity: We assessed our key performance indicators (see <u>APPENDIX B</u>) as completed or not completed to measure the extent to which each patient received each component of the CHICAGO Plan intervention, based on their allocation to the three treatment groups.
- (2) Focus groups: We completed debrief interviews with caregivers to better understand if they were satisfied with the content, comprehension, and relevance of the intervention material. We also asked about the satisfaction with the interventions provided by the ED coordinator and CHWs, and any other comments the patient or caregiver would like to offer about how to improve the CHICAGO Plan. We informed the participants that their responses would be used to help determine how to improve studies in the future (UIC IRB # 2017-0888).
- (3) Interviews of ED Coordinators, DCC Research Assistants, and CHWs: We asked study staff provide feedback about barriers and facilitators to completing study procedures (e.g., space or time constraints when providing ED-based instruction; availability of participants at scheduled home visit times). We informed study staff that their responses would be used to help determine how to improve studies in the future (UIC IRB # 2017-0888).

CHICAGO Plan Protocol 12-01-2017

#### XI. Timeline / milestones

366 367 368

369

370

We originally proposed a 15 month recruitment period, which was extended to be 18 months because of slow enrollment after approval by the Patient-Centered Outcomes Research institute. The planned date for end of the follow-up was also modified to allow the last enrolled participant to complete the 6-month follow-up assessment (primary endpoint).

371 372 373

#### Key dates

| | Original date | Final date (approved by study funder and DSMB) |
|---|---|---|
| Start of enrollment | March 1, 2015 | March 1, 2015 (no change) |
| End of enrollment period | May 31, 2016 | August 31, 2016 |
| End of study visits/data collection | November 30, 2016 | March 31, 2017 |

374

#### XII. Protection of human subjects

377378379

#### A. Risks to human subjects

380 381

382

383

384

385

386

Human subjects involvement and characteristics

The trial aimed to include approximately 640 children ages 5-11 years and their caregivers. The eligibility criteria are discussed in an earlier section of this protocol. Children and caregivers were randomly allocated to 1) ED-only; 2) ED-plus-home; or 3) Enhanced usual care. All participants were asked to complete study procedures for at least 6 months, regardless of the group they are assigned to; a study coordinator (masked to the treatment assignment) conducted assessment visits at baseline, 1, 3, and 6 months post index ED visit.

387 388

#### **B.** Sources of materials

389 390 391

392

393

Sources of materials included: Questionnaires administered by the ED coordinator (baseline data), and those administered by the DCC research assistant (follow-up data); Pharmacy dispensation data and electronic health records (EHR); Direct observation (e.g., home inspection / completion of environmental assessment checklist; review of inhaler technique using checklist).

394 395

#### C. Potential risk

396 397 398

399

400

401

402

403

404

405

406

407

408

409

410

411

412

Participants and caregivers were subject only to minimal risks through this research; we were testing two different approaches to promoting guideline recommended care (ED-only; ED-plushome) compared to usual Enhanced usual care. Potential risks included inconvenience or embarrassment involved in completing questionnaires or demonstrating self-management skills, or permitting the CHW (or research assistant) to conduct home visits for interventions (or for assessments), or in allowing the DCC to obtain pharmacy dispensation records (used for measuring adherence). The caregiver was not required to answer any questions (or conduct any part of the study) that he/she was reluctant to discuss/conduct. There was also a risk of loss of confidentiality. The CHW was instructed to avoid providing patients/caregivers with any type of medical advice, but had direct access to health care providers to address any patient/caregiver clinical questions or concerns. If the CHW was contacted about clinical questions, the CHW was instructed to connect the participant/caregiver with a health care provider familiar with the participant's medical condition immediately. On enrollment, caregivers were instructed to call their health care provider or seek emergency services in case of worsening symptoms, as opposed to directing questions to the CHW. All participants were informed in advance that they may withdraw from the study at any time without negatively affecting their medical care or any other benefits they might receive.

413 414 415

#### D. Adequacy of protection against risks

416 417

#### Recruitment and informed consent/assent

- We sought informed assent in all children that were capable of providing assent (age ≥7 years old) and permission of their caregiver in the ED. In children < 7 years old, consent was obtained from
- 420 the caregiver in the ED. As this study was no greater than minimal risk, the permission of only one
- 421 parent or guardian was sufficient for research to be conducted under the Additional Protections for
- Children Involved as Subjects in Research (45 CFR Part 46.404). Assent from the child and

permission or consent from the parent/guardian was be obtained by the ED coordinator at each participating clinical site. All staff were trained in informed consent/assent procedures and were available to read the consent/assent forms to individual with low literacy levels. The consent/assent forms were available in English and Spanish.

All caregiver/family information, including contact information, questionnaires, pharmacy dispensation and clinical information was available only available to designated members of the research team. Case report forms were locked in cabinets and electronic data was stored on password-protected files. Only authorized study staff had access to study data. Study reports presented to external collaborators did not contain any identifiable information and findings were presented in aggregate (or by treatment group).

#### <u>Incomplete disclosure</u>

As participants in this trial were aware of which treatment group they are assigned to, there was a risk for Hawthorne effect (change in behavior as a result of monitoring alone) and information bias as it relates to answering questions for the patient-reported outcomes (the primary outcomes and several secondary outcomes). Although there may have been changes in behavior (e.g., improved adherence to corticosteroids), our studies and those of others have shown that monitoring does not itself result in sustained adherence. To minimize this risk, however, there was incomplete disclosure of the interventions in the CHICAGO study during informed consent. The study was described as testing different communication strategies combining written and verbal instructions to all participants. Using doorknob hangers, as was successfully performed in a recent study, we aimed to mask the participants. Regardless of the arm the participant is randomized in, children and caregiver/families will receive a doorknob hanger in the form of a plasticized document, depicting one or more facts about asthma unrelated to the study interventions (e.g., recommendations for influenza vaccinations). To minimize the risk of bias, the DCC research assistant who collected outcome data was be masked to the treatment group.

Incomplete disclosure is generally necessary in studies of bias or social desirability (such as monitoring of adherence) and is considered acceptable by medical ethicists, the American Psychological Association, and IRBs when certain strict criteria are met. In designing this study, as with previous studies conducted by Dr. Krishnan, we had been guided by the American Psychological Association (APA) Ethics Code for conducting research. Specifically, we believed that incomplete disclosure was minimal risk to participants and was unavoidable since we were proposing to monitor behavior while minimizing the risk of Hawthorne effect. Moreover, we followed the recommendations of the APA and Bersoff et al. that call for a full debriefing of participants at the conclusion of the study.

#### E. Potential benefits of the proposed research to the subjects and others

It is difficult to know if the participants benefited from the research. All study participants/caregivers received instruction about appropriate MDI use with the teach-to-back methodology; they also received two MDI spacers for their use. Other than these specific benefits, we did not indicate any benefits from participating.

#### F. Importance of the knowledge to be gained

African American and Latino children suffer disproportionate asthma outcomes compared to non-Latino whites, as evidenced by emergency department (ED) visits for uncontrolled asthma. This study aimed to evaluate the effectiveness of using multi-level interventions to increase self-management skills and patient-centered outcomes in a minority pediatric ED population with uncontrolled asthma. If this intervention proves successful, it could make a significant impact in adherence to the asthma guidelines and equalize asthma care and health care utilization, among African American and Latino children with asthma. Risks to participants and their caregivers involved in the research were minimal.

#### G. Data safety monitoring plan

The study was reviewed by the IRB at each participating institution and approval was sought before study activities begin. We also submitted IRB continuing reviews annually and adverse event reports as specified by each IRB. This study used a Data and Safety Monitoring Board (DSMB) which included 5 individuals who were not affiliated with any of the participating institutions (1 chair with extensive expertise multi-center clinical trials, 2 pediatricians, 1 statistician, and 1 caregiver). The DSMB convened once in Year 1 (review/approve final study protocol) and twice per year in Year 2 and Year 3. The DSMB made affirmative decisions at each meeting whether to continue or terminate the study. Early termination was always an option for the DSMB, particularly if there were serious concerns about patient safety or there is evidence of futility or sufficient evidence of efficacy; decisions regarding early termination were made by the DSMB during convened meetings. No interim analyses of outcomes for efficacy or futility were planned before the study or requested by the DSMB throughout the study. In general, the DSMB was provided data grouped by treatment (i.e., masked to treatment assignment). If the DSMB had requested, for the purpose of competent deliberation, to see the treatment assignments (by group or individual), these would have been provided by the DCC biostatistician. Insofar as possible, the investigators remained masked to the treatment assignments of individual patients unless it was judged that it was in the best interests of an individual patient.

#### H. ClinicalTrials.gov requirements

This trial was registered in ClinicalTrials.gov prior to start of enrollment of participants. The results of the trial will be reported within the required timeframe. The registration will be updated and results be made available according to the requirements.

#### I. Inclusion of women and minorities

The proportion of girls included in the study intended to mirror the prevalence of this condition in the community and the patient population of the medical centers in which the study took place. The study took place at different medical centers that serve a large number of racial or ethnic minorities. The investigators anticipated that approximately 70% of participants would be African American, 15% Latino, 8% Caucasian and 7% other (Asian, Native American, Pacific Islander) reflecting the racial and ethnic background of our patient populations. Minorities were enrolled as they presented to enrollment sites, and Spanish-speaking participants were included.

#### XIII. References

- 1. U.S. Department of Health and Human Services (HHS). Expert panel report 3: Guidelines for the diagnosis and management of asthma. Bethesda, MD: HHS, National Heart, Lung and
- Blood Institute, National Institutes of Health. Publication No. 07–4051. 2007.
- http://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines (accessed November 30, 2017).
- Centers for Disease Control and Prevention: AsthmaStats.
   http://www.cdc.gov/asthma/asthma stats/ accessed November 30, 2017).
- Moorman JE, Akinbami LJ, Bailey CM, et al. National Surveillance of Asthma: United States,
   2001–2010. National Center for Health Statistics. Vital Health Stat 3(35). 2012.
- Akinbami LJ, Moorman JE, Simon AE, Schoendorf KC. Trends in racial disparities for
   asthma outcomes among children 0 to 17 years, 2001-2010. J Allergy Clin Immunol.2014
   Sep;134(3):547-553.
- 5. Illinois Department of Public Health. Asthma burden update, 2013.
- http://www.iedasp.org/iedasp/AsthmaBurdenBrief\_201305\_final.pdf accessed November 30, 2017).
- Cabana MD, Lara M, Shannon J. Racial and ethnic disparities in the quality of asthma care.
   Chest. 2007 Nov;132(5 Suppl):810S-817S.
- Crocker D, Brown C, Moolenaar R, Moorman J, Bailey C, Mannino D, Holguin F. Racial and ethnic disparities in asthma medication usage and health-care utilization: data from the National Asthma Survey. Chest. 2009 Oct;136(4):1063-71.
- 8. National Heart, Lung, and Blood Institute. National Asthma Education and Prevention Program Guidelines Implementation Panel Report.
- https://www.nhlbi.nih.gov/files/docs/guidelines/gip\_rpt.pdf accessed November 30, 2017).
  Weiss KB, Shannon JJ, Sadowski LS, Sharp LK, Curtis L, Lyttle CS, Kumar R, Shalowitz
- Weiss KB, Shannon JJ, Sadowski LS, Sharp LK, Curtis L, Lyttle CS, Kumar R, Shalowitz
   MU, Weiselberg L, Catrambone CD, Evans A, Kee R, Miller J, Kimmel L, Grammer LC. The
   burden of asthma in the Chicago community fifteen years after the availability of national
- asthma guidelines: the design and initial results from the CHIRAH study. Contemp Clin Trials. 2009; 30: 246-55.
- Shalowitz MU, Sadowski LM, Kumar R, Weiss KB, Shannon JJ. Asthma burden in a
   citywide, diverse sample of elementary school children in Chicago. Ambul Pediatr. 2007; 7:
   271-7.
- 11. Coordinated Healthcare Interventions for Childhood Asthma Gaps in Outcomes (CHICAGO)
   Plan. Respiratory Health Association. https://lungchicago.org/what-we-offer/research/collaborations/chicago-plan/ (accessed November 30, 2017).
- Krishnan JA, Schatz M, Apter AJ. A call for action: Comparative effectiveness research in
   asthma. J Allergy Clin Immunol. 2011 Jan; 127:123-7.
- 13. Lieu TA, Au D, Krishnan JA, Moss M, Selker H, Harabin A, Taggart V, Connors A; Comparative Effectiveness Research in Lung Diseases Workshop Panel. Comparative
- effectiveness research in lung diseases and sleep disorders: recommendations from the
- National Heart, Lung, and Blood Institute workshop. Am J Respir Crit Care Med. 2011 Oct 1;184(7):848-56.
- 14. Bender BG, Krishnan JA, Chambers DA, Cloutier MM, Riekert KA, Rand CS, Schatz M,
- Thomson CC, Wilson SR, Apter A, Carson SS, George M, Gerald JK, Gerald L, Goss CH,
- Okelo SO, Mularski RA, Nguyen HQ, Patel MR, Szefler SJ, Weiss CH, Wilson KC, Freemer

- M. American Thoracic Society and National Heart, Lung, and Blood Institute Implementation Research Workshop Report. Ann Am Thorac Soc. 2015 Dec;12(12):S213-21.
- Ducharme FM, Zemek RL, Chalut D, McGillivray D, Noya FJ, Resendes S, Khomenko L,
   Rouleau R, Zhang X. Written action plan in pediatric emergency room improves asthma
   prescribing, adherence, and control. Am J Respir Crit Care Med. 2011;183(2):195-203.
- Krieger JW, Takaro TK, Song L, Weaver M. The Seattle-King County Healthy Homes
   Project: A randomized, controlled trial of a community health worker intervention to decrease
   exposure to indoor asthma triggers. Am J Public Health 2005; 95: 652-9.
- Krieger J, Takaro TK, Song L, Beaudet N, Edwards K. A randomized controlled trial of
   asthma self-management support comparing clinic-based nurses and in-home community
   health workers: The Seattle-King County Healthy Homes II Project. Arch Pediatr Adolesc
   Med. 2009; 163: 141-9.
- 18. Crocker DD, Kinyota S, Dumitru GG, Ligon CB, Herman EJ, Ferdinands JM, Hopkins DP, Lawrence BM, Sipe TA; Task Force on Community Preventive Services. Effectiveness of home-based, multi-trigger, multicomponent interventions with an environmental focus for reducing asthma morbidity: a community guide systematic review. Am J Prev Med. 2011 Aug;41(2 Suppl 1):S5-32.
- 19. Nurmagambetov TA, Barnett SB, Jacob V, Chattopadhyay SK, Hopkins DP, Crocker DD, Dumitru GG, Kinyota S; Task Force on Community Preventive Services. Economic value of home-based, multi-trigger, multicomponent interventions with an environmental focus for reducing asthma morbidity a community guide systematic review. Am J Prev Med. 2011 Aug;41(2 Suppl 1):S33-47.
- 20. Patient Centered Outcomes Research Institute.
   https://www.pcori.org/sites/default/files/PCORI-PFA-Asthma-061813.pdf (accessed
   November 30, 2017).
- Martin MA, Press VG, Nyenhuis SM, Krishnan JA, Erwin K, Mosnaim G, Margellos-Anast
   H, Paik SM, Ignoffo S, McDermott M; CHICAGO Plan Consortium. Care transition
   interventions for children with asthma in the emergency department. J Allergy Clin Immunol.
   2016;138(6):1518-1525.
- Erwin K, Martin MA, Flippin T, Norell S, Shadlyn A, Yang J, Falco P, Rivera J, Ignoffo S,
   Kumar R, Margellos-Anast H, McDermott M, McMahon K, Mosnaim G, Nyenhuis SM, Press
   VG, Ramsay JE, Soyemi K, Thompson TM, Krishnan JA. Engaging stakeholders to design a
   comparative effectiveness trial in children with uncontrolled asthma. J Comp Eff Res 2016; 5:
   17-30.
- Martin MA, Press VG, Erwin K, Margellos-Anast H, Ignoffo S, McMahon KS, Mosnaim G,
   Ramsay J, Paik SM; CHICAGO Plan Investigators. Engaging end-users in intervention
   research study design. J Asthma. 2017:1-9.
- Erwin K, Norell S, Martin MA, Paik M, Press VG, Thompson TA, Krishnan JA. Applying design methods to care delivery science: Improving the care of minority children with uncontrolled asthma and their caregivers who present to six Emergency Departments in Chicago through a stakeholder-optimized discharge tool. Journal of Information Design 2017 (accepted, in press).
- Krishnan JA, Martin MA, Lohff C, Mosnaim GS, Margellos-Anast H, DeLisa JA, McMahon
   K, Erwin K, Zun LS, Berbaum ML, McDermott M, Bracken NE, Kumar R, Margaret Paik S,
   Nyenhuis SM, Ignoffo S, Press VG, Pittsenbarger ZE, Thompson TM; CHICAGO Plan
   consortium. Design of a pragmatic trial in minority children presenting to the emergency

- department with uncontrolled asthma: The CHICAGO Plan. Contemp Clin Trials. 2017 Jun; 57:10-22.
- Yancey AK, Ortega AN, Kumanyika SK. Effective recruitment and retention of minority
   research participants. Annu Rev Public Health. 2006; 27: 1-28.
- Nicholson LM, Schwirian PM, Klein EG, Skybo T, Murray-Johnson L, Eneli I, Boettner B,
   French GM, Groner JA. Recruitment and retention strategies in longitudinal clinical studies
   with low-income populations. Contemp Clin Trials 2011; 32: 353-62.
- 28. Bersoff DM, Bersoff DN. Ethics and self-report data. In: Stone A, Turkkan JS, Bachrach
   CA, Jobe JB, Kurtzman HS, Cain VS, eds. The science of self-report: implications for
   research and practice. Mahwah, NJ: Lawrence Erlbaum Associates, 1999: 9-24
- 29. American Psychological Association. Ethical principles of psychologists and code of conduct. Am Psychol 1992; 47: 1597-1611.
- 30. Rochon, J. Sample size calculations for two-group repeated-measures experiments. Biometrics 1991, 47:1383–1398.
- 619 31. Cohen, J. Statistical power analysis for the social sciences. 2nd ed. New York: Routledge; 620 1988.
- Health measures: meaningful change. http://www.healthmeasures.net/score-and-interpret/interpret-scores/meaningful-change. (accessed November 30, 2017)
- 33. Thissen D, Liu Y, Magnus B, Quinn H, Gipson DS, Dampier C, Huang IC, Hinds PS,
   Selewski DT, Reeve BB, Gross HE, DeWalt DA. Estimating minimally important difference
   (MID) in PROMIS pediatric measures using the scale-judgment method. Qual Life Res.
   2016;25: 13-23.
- 34. Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92.
- 35. Press VG, Arora VM, Shah LM, Lewis SL, Ivy K, Charbeneau J, Badlani S, Nareckas E,
   Mazurek A, Krishnan JA. Misuse of respiratory inhalers in hospitalized patients with asthma
   or COPD. J Gen Intern Med 2011; 26: 635-42.
- 36. Press VG, Arora VM, Trela KC, Adhikari R, Zadravecz FJ, Liao C, Naureckas E, White SR,
   Meltzer DO, Krishnan JA. Effectiveness of Interventions to Teach Metered-Dose and Diskus
   Inhaler Techniques. A Randomized Trial. Ann Am Thorac Soc 2016; 13: 816-24.
- Okelo SO, Butz AM, Sharma R, Diette GB, Pitts SI, King TM, Linn ST, Reuben M,
   Chelladurai Y, Robinson KA. Interventions to modify health care provider adherence to
   asthma guidelines: a systematic review. Pediatrics 2013; 132: 517-34.
- 38. Health Measures: Transforming How Health Is Measured. Patient Reported Outcomes
   Measurement Information System (PROMIS).
- http://www.healthmeasures.net/exploremeasurement-systems/promis (accessed November 30, 2017).
- 39. Patient-Reported Outcomes Measurement Information System. Dynamic Tools to Measure
   Health Outcomes From the Patient Perspective: Asthma Impact.
- https://www.assessmentcenter.net/documents/PROMIS%20Asthma%20Impact%20Scoring% 20Manual.pdf (accessed November, 28 2017)
- 40. Howell CR, Thompson LA, Gross HE, Reeve BB, DeWalt DA, Huang IC. Responsiveness to
   Change in PROMIS Measures among Children with Asthma: A Report from the PROMIS
   Pediatric Asthma Study. Value Health. 2016; 19: 192-201.

- 41. Patient-Reported Outcomes Measurement Information System. Dynamic Tools to Measure
   Health Outcomes From the Patient Perspective: Satisfaction with Participation in Social
   Roles.
- https://www.assessmentcenter.net/documents/PROMIS%20[Satisfaction%20with%20Particip ation%20in%20Social%20Roles]%20Scoring%20Manual.pdf (accessed November, 30 2017)
- Hahn EA, Beaumont JL, Pilkonis PA, Garcia SF, Magasi S, DeWalt DA, Cella D. The
   PROMIS satisfaction with social participation measures demonstrated responsiveness in
   diverse clinical populations. J Clin Epidemiol 2016; 73: 135-41.
- Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R.
   Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy
   Clin Immunol 2007 Apr;119(4):817-25.
- 44. Bime C, Gerald JK, Wei CY, Holbrook JT, Teague WG, Wise RA, Gerald LB. Measurement
   characteristics of the childhood Asthma-Control Test and a shortened, child-only version. NPJ
   Prim Care Respir Med. 2016 Oct;26:16075.
- Liu AH, Zeiger RS, Sorkness CA, Ostrom NK, Chipps BE, Rosa K, Watson ME, Kaplan MS,
   Meurer JR, Mahr TA, Blaiss MS, Piault-Louis E, McDonald J. The Childhood Asthma
   Control Test: retrospective determination and clinical validation of a cut point to identify
   children with very poorly controlled asthma. J Allergy Clin Immunol. 2010 Aug;126(2):267 73.
- 46. Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009
   Oct;124(4):719-23.
- 47. Akinbami LJ, Sullivan SD, Campbell JD, Grundmeier RW, Hartert TV, Lee TA, Smith RA.
   Asthma outcomes: healthcare utilization and costs. J Allergy Clin Immunol. 2012 Mar;129(3
   Suppl):S49-64.
- 48. Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in children with asthma. Quality of Life Research 1995 May; 5:35-46.
- 49. Stelmach I, Podlecka D, Smejda K, Majak P, Jerzyńska J, Stelmach R, Janas A, Stelmach W.
   Pediatric asthma caregiver's quality of life questionnaire is a useful tool for monitoring asthma in children. Qual Life Res 2012; 21:1639-42.
- 50. American Thoracic Society: Quality of Life Resource. Pediatric Asthma Caregiver's Quality of Life Questionnaire. http://qol.thoracic.org/sections/instruments/pt/pages/pacqlq.html (accessed November, 30 2017)
- 51. Patient-Reported Outcomes Measurement Information System. Dynamic Tools to Measure
   Health Outcomes From the Patient Perspective: Anxiety.
- https://www.assessmentcenter.net/documents/PROMIS%20Anxiety%20Scoring%20Manual.p df (accessed November, 30 2017)
- 52. Patient-Reported Outcomes Measurement Information System. Dynamic Tools to Measure
   Health Outcomes From the Patient Perspective: Depression.
- https://www.assessmentcenter.net/documents/PROMIS%20Depression%20Scoring%20Manu al.pdf (accessed November, 30 2017).
- 53. Patient-Reported Outcomes Measurement Information System. Dynamic Tools to Measure Health Outcomes From the Patient Perspective: Fatigue.
- https://www.assessmentcenter.net/documents/PROMIS%20Fatigue%20Scoring%20Manual.p df (accessed November, 30 2017)

- 54. Patient-Reported Outcomes Measurement Information System. Dynamic Tools to Measure
   Health Outcomes From the Patient Perspective: Sleep Disturbance.
- https://www.assessmentcenter.net/documents/PROMIS%20Sleep%20Disturbance%20Scoring %20Manual.pdf (accessed November, 30 2017)
- 55. National Institutes of Health / National Heart, Lung, and Blood Institute. National Asthma
   Education and Prevention Program. Guidelines for the Diagnosis and Management of Asthma
   (EPR-3). https://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines
   (accessed November, 30 2017)
- Hasegawa K, Sullivan AF, Tsugawa Y, Turner SJ, Massaro S, Clark S, Tsai CL, Camargo CA
   Jr; MARC-36 Investigators. Comparison of US emergency department acute asthma care
   quality: 1997-2001 and 2011-2012. J Allergy Clin Immunol. 2015 Jan;135(1):73-80.
- 57. Hedeker D, Gibbons RD. Longitudinal data analysis. Hoboken, NJ: John Wiley & Sons,
   Inc., 2006.
- 58. Li P, Stuart EA, Allison DB. Multiple Imputation: A Flexible Tool for Handling Missing Data. JAMA. 2015;314(18):1966-1967.
- 59. Li Y, De A. Multiple imputation by fully conditional specification for dealing with missing data in a large epidemiologic study. Int J Stat Med Res 2015; 4(3): 287-295.
- 712 60. Anise A, Hasnain-Wynia R. Patient-centered outcomes research to improve asthma outcomes.
   713 J Allergy Clin Immunol. 2016 Dec;138(6):1503-1510.
- 714 61. Illinois Department of Public Health. Illinois Asthma State
  715 Planhttp://www.dph.illinois.gov/sites/default/files/publications/publicationsohpmillinois716 asthma-state-plan.pdf (accessed November 30, 2017)

718 XIV. Appendices

719 720

721 A. CAPE tool

722 B. Key performance indicators

723

# APPENDIX A1. CAPE -Asthma Discharge Plan (Version June 19, 2015)

| | | discharge plan | Child's name Today's date Doctor's signature | |
|---|---|---|---|---|
| Your ora<br>steroid i | Liquid | 1st dose time/date | Things to know about oral steroids: • is another powerful "rescue" medicine • if you were given these in the emergency room, it is very important that you finish them! | |
| Your "remedicin | scue" e is: Spacer Nebulizer | 1st dose time/date | with symptoms | Mark your meds<br>at the pharmacy:<br>red sticker for<br>"rescue"<br>medicine |
| Your "co<br>medicin<br>Inhaler<br>Mask | ntroller" e is: Spacer Nebulizer | 1st dose time/date | Things to know about controller medicine: • should be used every day, even if your child has no symptoms • examples include Pulmicort, Flovent, Azmacort, Advair • may be an allergy medication, such as Singulair and Accolate | Mark your meds at the pharmacy: (green sticker for "controller" medicine |
| | See your | child's doctor within 3 days o | f your ER visit | |



# Read the signs





# Stay on top of asthma

Don't wait! Call with questions

**Call your child's regular doctor as soon as possible** to help you understand your child's asthma and home treatment plan.

ldentify your child's asthma triggers

**Build a trigger list** of what seems to make your child's asthma act up. Add to that list as you notice new triggers. Try to help your child avoid these!

**If your child has a cold**, use your child's action plan; and help them to blow their nose.

**Avoid smoking**—a known asthma trigger—and avoid having your child in a house where someone smokes.

Here are some examples of common asthma triggers:













| What are your child's triggers | ? |
|--------------------------------|---|

| | Give |
|---|---------------|
| - | medications |
| | as proscribed |

**Review how to use** the inhalers with your child's doctor. **Develop tricks** to help remind you to give the medications.

| What might be useful tricks? | |
|------------------------------|----------------------------------|
| 3 | set an alert on your smartphone |
| | keep medicine by your coffee pot |

Take your child to the doctor regularly

**Your child's doctor is there to help**—they want to see how well your child is doing and to review your child's symptom control.

Together you and your doctor will discuss a new Asthma Home Plan, with instructions for when your child's asthma is under control and when it is not well-controlled.



## How to use an inhaler with a spacer

Works as well as a nebulizer!



Take cap off the inhaler. Check for and remove any dust, lint, or other objects. Shake the inhaler well.



Attach the inhaler to the spacer.



Breathe out all the air, away from the spacer.



Put lips around device, press inhaler one time. This puts one puff of medicine into the spacer.



Breathe in deeply and slowly, and hold your breath.



**Remove** the device from the mouth. Then **hold** your breath for 5 secs. Then breathe normally **away** from the spacer.



If your child needs to take another puff of medicine, wait 1 minute. After one minute, repeat steps 3 to 6.



Rinsing is only necessary if the medicine you just took was an inhaled steroid. Have your child rinse his or her mouth out with water after the last puff of medicine. **Make sure your child spits the water out.** Do not allow the child to swallow the water. Recap the inhaler.

From the American College of Chest Physicians Ilustrations by Paula Falco

© 2015 CHICAGO Plan Investigators + PCORI The CHICAGO Plan is a PCORI-funded study comparing asthma interventions. For questions regarding this document or the CHICAGO Plan, contact: Trevonne Thompson, MD, tthomps@uic.edu



**What is this?** This is a QR code. To use it, go to the app store on your smartphone, search for 'QR code readers' and download the free app.

To learn more about asthma, scan this code with the app to link to the Respiratory Health Association website. Or go to the link below: www.tinyurl.com/asthmalib

| | | home plan | Child's name Today's date Doctor's signature | Date |
|---|---|---|---|---|
| Your "comedicin Inhaler Mask | ontroller" e is: Spacer Nebulizer | Number of puffs How often Take every day EVEN IF no visible symptoms | Things to know: • should be used every day, even if your child has no symptoms • examples include Pulmicort, Flovent, Azmacort, Advair • may be an allergy medication, such as Singulair and Accolate | Mark your meds at the pharmacy: (green sticker for "controller" medicine |
| Your "remedicin | | Number of puffs How often Use when symptoms occur Use 5 - 15 minutes before exercise | Things to know: • should be used only if your child is having symptoms during an asthma attack/ with symptoms • is typically albuterol with a name like: Proventil, Pro-Air, Ventolin, Xopenex | Mark your meds at the pharmacy: red sticker for "rescue" medicine |
| Other: | | | | |



# See your child's doctor regularly

Doctor's name and phone number

Next appointment date and time

# Read the signs







743 744



# Stay on top of asthma

Don't wait! Call with questions

**Call your child's regular doctor** with any questions about how to use your child's Asthma Home Plan.

ldentify your child's asthma triggers

**Build a trigger list** of what seems to make your child's asthma act up. Add to the list as you notice new triggers. Try to help your child avoid these!

**If your child has a cold**, use your child's action plan; and help them to blow their nose.

**Avoid smoking**—a known asthma trigger—and avoid having your child in a house where someone smokes.

Here are some examples of common asthma triggers:



| What are your child's triggers? |
|---------------------------------|

Give medications as prescribed

**Review how to use** the inhalers with your child's doctor.

**Develop tricks** to help remind you to give the medications.

| What might be useful tricks? | |
|------------------------------|----------------------------------|
| 3 | set an alert on your smartphone |
| | keep medicine by your coffee pot |

Take your child to the doctor regularly

**Your child's doctor is there to help**—they want to see how well your child is doing and to review your child's symptom control.

Together you and your doctor will talk about your Asthma Home Plan. Your doctor will make changes to the plan to help you stay on top of your child's asthma.



# How to use an inhaler with a spacer

#### Works as well as a nebulizer!



Take cap off the inhaler. Check for and remove any dust, lint, or other objects. Shake the inhaler well.



Attach the inhaler to the spacer.



Breathe out all the air, away from the spacer.



Put lips around device, press inhaler one time. This puts one puff of medicine into the spacer.



Breathe in deeply and slowly, and hold your breath.



Remove the device from the mouth. Then hold your breath for 5 secs. Then breathe normally away from the spacer.



If your child needs to take another puff of medicine, wait 1 minute. After one minute, repeat steps 3 to 6.



Rinsing is only necessary if the medicine you just took was an inhaled steroid. Have your child rinse his or her mouth out with water after the last puff of medicine. Make sure your child spits the water out. Do not allow the child to swallow the water. Recap the inhaler.

© 2015 CHICAGO Plan Investigators + PCORI The CHICAGO Plan is a PCORI-funded study

comparing asthma interventions. For questions regarding this document or the CHICAGO Plan, contact: Trevonne Thompson, MD, tthomps@uic.edu



What is this? This is a QR code. To use it, go to the app store on your smartphone, search for 'QR code readers' and download the free app.

To learn more about asthma, scan this code with the app to link to the Respiratory Health Association website. Or go to the link below: www.tinyurl.com/asthmalib



From the American College of Chest Physicians Ilustrations by Paula Falco

| /52 | APPE | INDIX B: Key performance indicators |
|---|---|---|
| 753<br>754 | | ach, we will monitor the % completion on a monthly basis at our Steering Committee meetings rovide these key performance metrics to the DSMB prior to the scheduled meetings. |
| 755 | | |
| 756 | A. En | nergency Department (ED)-level intervention performance metrics |
| 757 | | |
| 758<br>759 | (1) | Randomize n children/caregivers per month per site X 15 months (hereafter referred to as participants). The per-site n values are based on historical data from each site: |
| 760 | | A. John H. Stroger Jr. Hospital of Cook County: 1.7 children/caregivers per month |
| 761 | | B. Lurie Children's Hospital of Chicago: 17.5 children/caregivers per month |
| 762 | | C. Rush University Medical Center: 3.9 children/caregivers per month |
| 763 | | D. Sinai Health System: 4.0 children/caregivers per month |
| 764 | | E. University of Chicago: 12.7 children/caregivers per month |
| 765<br>766 | | F. University of Illinois Hospital & Health Sciences System/University of Illinois at Chicago: 2.6 children/caregivers per month |
| 767 | (2) | % of participants who meet study eligibility criteria |
| 768<br>769<br>770 | (3) | % of participants who have appropriate documentation of informed consent (written informed consent and assent) Age that assent is needed varies by site, listed below (site: age for assent): |
| 771 | | A. John H. Stroger Jr. Hospital of Cook County: 7 years old |
| 772 | | B. Lurie Children's Hospital of Chicago: 12 years old |
| 773 | | C. Rush University Medical Center: 8 years old |
| 774 | | D. Sinai Health System: 8 years old |
| 775 | | E. University of Chicago: 8 years old |
| 776<br>777 | | F. University of Illinois Hospital & Health Sciences System/University of Illinois at Chicago: 7 years old |
| 778<br>779<br>780<br>781<br>782<br>783 | (4) | % of participants who receive the intervention as per randomized treatment assignment: (a) for the Usual Care group, the ED coordinator provides MDI instruction and Doorknob hanger; (b) for CAPE group, ED coordinator provides MDI instructions, Doorknob hanger, and completes the CAPE with the participants prior to ED discharge; (c) for ED-plus-home group, ED coordinator provides MDI instructions, Doorknob hanger, completes the CAPE with the participants prior to ED discharge, and arranges appointment for the first home visit by the community health worker. |

| 785 | | |
|---|---|---|
| 786<br>787 | Additional ED-level performance indicators for participants assigned to CAPE groups (ED-only or ED-plus-home): | |
| 788 | | |
| 789<br>790<br>791 | (5) | % of participants who were prescribed a systemic corticosteroid for use after ED discharge (as measured by documentation of a new prescription, an active prescription, or other instructions to use systemic corticosteroids after discharge.) |
| 792<br>793<br>794<br>795 | (6) | % of participants who) were prescribed inhaled corticosteroids (or another controller) for use after ED discharge (as measured by documentation of a new prescription, an active prescription, or other instructions to use inhaled corticosteroids or another controller after discharge) |
| 796<br>797 | (7) | % of participants who received a post-ED follow-up appointment with the child's provider within 28 days of ED discharge (date/time/name), |
| 798<br>799<br>800 | (8) | % of participants who were prescribed a rescue /quick-relief medication for use after ED discharge (as measured by documentation of a new prescription, an active prescription, or other instructions to use a rescue/quick-relief medication after discharge) |
| 801<br>802<br>803 | (9) | % of participants who received instruction using teach-to-goal methodology to (a) increase comprehension about (5) to (8), (b) green/yellow/red zones of the asthma action plan, and (c) need to avoid known environmental triggers; |
| 804 | | |
| 805<br>806<br>807<br>808 | study<br>evalua | te project manager will conduct ED chart reviews within 3-4 business days of discharge for all participants to assess (5) to (9). These data will be used to assess performance and to also atte the extent to which there is contamination across treatment groups. Training or re-training e performed and documented on a case-by-case basis. |
| 809 | | |
| 810<br>811 | B. Ho home | me visit-level intervention performance metrics (for participants randomized to ED-plus- |
| 812 | | |
| 813<br>814<br>815 | consid | rmance metrics for completion of home visits by community health worker (CHW). We will der 3 levels of completion: within window, after window has ended, and not completed for the ving metrics: |
| 816<br>817 | (10) | % of participants who receive Home Visit #1 within 3 business days of discharge (window ends 3 business days after discharge) |
| 818<br>819 | (11) | % of participants who receive Home Visit #2 within 17 calendar days of discharge (window is 14 days +/- 3 calendar days) |

CHICAGO Plan Protocol 12-01-2017

- 820 (12) % of participants who receive Home Visit #3 within 37 calendar days of discharge (window is 30 days +/- 7 calendar days)
- % of participants who receive Home Visit #4 within 97 calendar days of discharge (window is 90 days +/- 7 calendar days)
- 824 (14) % of participants who receive Home Visit #5 within 187 calendar days of discharge (window is 180 days +/- 7 calendar days)

- Performance metrics for completion of all elements of each home visit:
- % of participants who receive each of the following elements by the CHW during Home Visit #1: introduction and explanation of the CHICAGO Plan; review asthma action plan developed in ED (CAPE); review of asthma basics; review of symptom recognition and understanding of controlled (green zone) vs. uncontrolled asthma (yellow/red zones): teachto-goal instruction about use of MDIs; assistance to develop a behavior change plan (related to preceding elements)
- % of participants who receive each of the following elements by the CHW during Home 834 (16)Visit #2: review asthma action plan updated since ED discharge in collaboration with 835 patient's provider (CAPE); review of asthma basics; review of symptom recognition and 836 understanding of controlled (green zone) vs. uncontrolled asthma (yellow/red zones): teach-837 to-goal instruction about use of MDIs; identification of and help with strategies to reduce the 838 3 major triggers; assess progress towards behavior change plan developed during home visit 839 #1 and assistance to develop updated plan (related to preceding elements); educate about 504 840 plan and how to submit paperwork (school nursing and administrative support) 841
- % of participants who receive each of the following elements by the CHW during Home Visit #3: review asthma action plan updated since ED discharge in collaboration with patient's provider (CAPE); teach-to-goal instruction about use of MDIs; identification of and help with strategies to reduce the 3 major triggers; assess progress towards behavior change plan developed during home visit #2 and assistance to develop updated plan (related to preceding elements); educate about 504 plan and how to submit paperwork (school nursing and administrative support)
- % of participants who receive each of the following elements by the CHW during Home
  Visit #4: review asthma action plan updated since ED discharge in collaboration with
  patient's provider (CAPE); teach-to-goal instruction about use of MDIs; identification of and
  help with strategies to reduce the 3 major triggers; assess progress towards behavior change
  plan developed during home visit #3 and assistance to develop updated plan (related to
  preceding elements); educate about 504 plan and how to submit paperwork (school nursing
  and administrative support)

% of participants who receive each of the following elements by the CHW during Home 856 (19)Visit #5: review asthma action plan updated since ED discharge in collaboration with 857 patient's provider (CAPE); teach-to-goal instruction about use of MDIs; identification of and 858 help with strategies to reduce the 3 major triggers; assess progress towards behavior change 859 860 plan developed during home visit #4 and assistance to develop updated plan (related to preceding elements); educate about 504 plan and how to submit paperwork (school nursing 861 and administrative support). 862 863 The Data Coordinating Center collected these data in the REDcap database, which was used by the 864 CHW to document attempted and completed home visits. The Supervising CHWs (from the Sinai 865 CHW Coordinator Center) accompanied CHWs during home visits in a sample of home visits to 866 review in-person site-specific CHW performance. Training or re-training was performed and 867 868 documented on a case-by-case basis. 869 C. DCC data collection performance metrics (for all participants) 870 Performance metrics for data collection. We considered 3 levels of completion: within window, after 871 window has ended, and not completed for the following metrics: 872 873 % of participants with in-person BASELINE data collection prior to ED discharge 874 (20)% of participants with 1-month FOLLOW-UP data within 52 calendar days of discharge (21) 875 (window is 38 days + 14 calendar days) 876 % of participants with 3-month FOLLOW-UP data within 112 calendar days of discharge 877 (22)(window is 98 days + 14 calendar days) 878 % of participants with 6-month FOLLOW-UP data within 202 calendar days of discharge (23)879 (window is 188 days + 14 calendar days) 880 % of participants with 12-month FOLLOW-UP data within 367 calendar days of discharge (24)881 (window is 360 days +/- 7 calendar days); this data collection time-point is only for those 882 participants enrolled within first 7.5 months of enrollment period (50% of enrollment period) 883 to ensure there is adequate observation time for data collection at 12 months. 884 885 During the conduct of the study, we reviewed missing data and time to complete data collection; these data were used to provide feedback and additional training to study staff as needed. 886 The Data Coordinating Center collected these data in the REDcap database, which will be used by 887

the DCC research assistants to document attempted and completed outcome assessments. Training or

re-training was performed and documented on a case-by-case basis.

888

The study design employed the "large simple trial" or "pragmatic trial" format, rather than an efficacy design. The target performance varied by metric. For elements linked to human subjects protection (e.g., obtaining written informed consent from the caregiver; assent from the child >7yrs), the definition for major protocol deviation is <100%. For elements linked to implementing the interventions or data collection linked to specific time points, the definition for major protocol deviation is <50%. The goal is 100% performance on all metrics; we will ask site PIs to develop a written corrective action plan if site-level performance for implementing the protocol is <80% (<100% if there are deviations linked to human subjects protection). We reported major protocol deviations to the DSMB within 14 days after the event has been discovered by the contact PI. Depending on the site-specific reporting requirements, we may also report major deviations to the site's Institutional Review Board (IRB); for example, we will report all instances where informed consent was not obtained, but, depending on the institution may not need to report completion rates of study visits prior to the annual continuing review date for that institution's IRB.